CLINICAL TRIAL: NCT01551134
Title: IS Laparoscopic Fundoplication Superior to Open Fundoplication in Children - a Randomized Study
Brief Title: Is Laparoscopic Fundoplication Better Than Open Fundoplication in Children ?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Fewer patients than anticipated were referred
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-03082
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Fundoplication; Randomized Controlled Trial; General Surgery; Child; Laparoscopy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open fundoplication (Active Comparator): Fundoplication performed with open surgery
  Interventions: Procedure: Fundoplication
- Lap fundoplication (Experimental): Primary fundoplication performed by laparoscopic surgery
  Interventions: Procedure: Fundoplication

INTERVENTIONS:
Procedure: Fundoplication — Primary fundoplication
  Other Names: Gastroesophageal reflux
  Arms: Open fundoplication
Procedure: Fundoplication — Primary fundoplication
  Other Names: Gastroesophageal reflux
  Arms: Lap fundoplication

SUMMARY:
The aim of the study was to compare short- and longterm outcomes after laparoscopic and open Nissen fundoplication in children.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-15 years
* All patients accepted for primary fundoplication at Oslo University Hospital

Exclusion Criteria:

* Age over 16 years
* Parents not speaking Norwegian or English well
* Prior fundoplication
* Patients with comorbidities considered as unsuited for laparoscopic surgery (diaphragma hernia, several previous abdominal operations etc)

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2003-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Recurrence of reflux | 12, 24 and 48 months
  GER symptoms and GER on pH monitoring. Need for redo fundoplication. PPI.

SECONDARY OUTCOMES:
Postoperative complication rate | 30 days
  Perioperative complications. Duration of surgery. Postoperative complications. Lenght of hospital stay. Readmission to hospital.
Inflammatory response | The first 4 p.o days
  indicies of inflammatory response
Parental stress | 12 and 24 months
  Indicies of parental stress caused by GER pre- and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bjornland, MD, PhD, Principal Investigator — Department of hepatic, gastrointestinal and pediatric surgery, Oslo University Hospital HF, Rikshospitalet, Postboks 4950 Nydalen, 0424 Oslo, NORWAY.
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Fyhn TJ, Kvello M, Edwin B, Schistad O, Pripp AH, Emblem R, Knatten CK, Bjornland K. Outcome a decade after laparoscopic and open Nissen fundoplication in children: results from a randomized controlled trial. Surg Endosc. 2023 Jan;37(1):189-199. doi: 10.1007/s00464-022-09458-6. Epub 2022 Aug 1. PMID 35915187
- [Derived] Kvello M, Avitsland TL, Knatten CK, Fyhn TJ, Malt U, Emblem R, Bjornland K. Psychologic Distress and Anxiety in Mothers of Children With Gastroesophageal Reflux Undergoing Antireflux Surgery. J Pediatr Gastroenterol Nutr. 2019 Jun;68(6):818-823. doi: 10.1097/MPG.0000000000002286. PMID 31124989